CLINICAL TRIAL: NCT06767527
Title: A Randomized, Controlled, Multi-center Phase III Clinical Study of AK112 Plus Nab-paclitaxel Versus Placebo Plus Nab-paclitaxel as First-line Treatment for Locally Advanced Unresectable or Metastatic Triple-negative Breast Cancer
Brief Title: AK112 or Placebo Plus Nab-Paclitaxel as First-line Treatment in Inoperable Locally Advanced/ Metastatic Triple-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-308
Record Dates: First submitted 2025-01-08; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Triple-Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 (Experimental): AK112 Plus Nab-Paclitaxel
  Interventions: Drug: AK112; Drug: Nab-paclitaxel
- Placebo (Placebo Comparator): Placebo Plus Nab-Paclitaxel
  Interventions: Drug: Nab-paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: AK112 — AK112 via intravenous (IV) infusion
  Arms: AK112
Drug: Nab-paclitaxel — Nab-Paclitaxel 100mg/m2 via IV infusion on Days 1, 8, and 15 of each 28-day cycle
Drug: Placebo — Placebo via IV infusion
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind study aims to assess the safety and efficacy of AK112 in combination with Nab-Paclitaxel, compared to a placebo plus Nab-Paclitaxel, as a first-line treatment for inoperable locally advanced or metastatic triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form.
2. Age at enrollment is ≥ 18 and ≤ 75 years, both males and females are eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 3 months.
5. Histologically confirmed unresectable locally advanced or metastatic breast cancer with negative status for ER, PR, and HER-2.
6. Subjects who have not received prior systemic treatment for advanced breast cancer are eligible for the study.
7. Suitable for monotherapy with taxane-based agents.
8. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
9. Adequate organ function.

Exclusion Criteria:

1. Patients with locally recurrent disease who are eligible for surgery or radiotherapy.
2. History of other malignancies within the past 5 years.
3. Active autoimmune disease requiring systemic treatment within the past 2 years.
4. Pregnant or breastfeeding women.
5. Concurrent participation in another clinical trial, unless it is an observational or non-interventional study or in the follow-up phase of an interventional study.
6. Participants with clinically symptomatic pleural effusion, pericardial effusion, or ascites that require repeated drainage.
7. Participants with a history of immune deficiency; those who test positive for HIV antibodies; those currently using systemic corticosteroids or other immunosuppressive agents on a long-term basis.
8. Individuals with known active tuberculosis (TB), or those suspected of having active TB (who must undergo clinical evaluation for exclusion), and those with known active syphilis infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRRC | Up to approximately 2 years
  Progression-Free Survival (PFS) assessed by Independent Radiologic Review Committee (IRRC)
OS | Up to approximately 4 years
  Overall survival (OS) is defined as the time from randomization to death due to any cause

SECONDARY OUTCOMES:
PFS assessed by investigator | Up to approximately 2 years
  Progression-free survival is defined as the time from randomization to the first documented PD per RECIST 1.1 based on assessments by investigator or death due to any cause, whichever occurs first.
ORR assessed by IRRC or investigators | Up to approximately 2 years
  Objective Response Rate (ORR) is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experienced a CR or PR as assessed by IRRC or investigators based on RECIST 1.1 is presented.
DCR assessed by IRRC or investigators | Up to approximately 2 years
  Disease control rate (DCR) is defined as the sum rate of CR, PR and Stable Disease (SD), as determined by IRRC or investigators using RECIST v1.1
DoR assessed by IRRC or investigators | Up to approximately 2 years
  Duration of response (DoR) is defined as the time period from the date of initial CR or PR until the date of PD or death due to any cause, whichever occurs first.
TTR assessed by IRRC or investigators | Up to approximately 2 years
  Time to response (TTR) is defined as the time to response based on RECIST v1.1.
Adverse Events (AEs) | Up to approximately 2 years
  Incidence and severity of participants with adverse events
Cmax and Cmin | Up to approximately 2 years
  AK112 serum drug concentrations in subjects at different time points after AK112 administration.
Anti-drug antibodies (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China